CLINICAL TRIAL: NCT04579029
Title: Prospective Randomized Evaluation of Lymphaticovenous Anastomosis Using Dynamic Imaging in Breast Cancer-related Lymphoedema
Brief Title: PRELUDE Study of Lymphatic Surgery to Treat Breast Cancer Related Lymphoedema
Acronym: PRELUDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR4772
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical Cohort (Experimental): Patients randomised to the surgical group will undergo near infrared spectroscopy imaging to assess suitability and plan the surgical procedure.
  Limb measurements with perometry and bio-impedance spectroscopy will be performed at baseline. Under general anaesthetic multiple LVA bypass procedures will be performed on the affected arm. Near infrared spectroscopy imaging will be used throughout. One week after discharge the patient will return for the bandages to be removed and the wounds inspected for any evidence of infection before renewing the bandage. Again, two weeks after surgery, the patient will return for inspection of wound and removal of sutures. It is at this point that the surgical patients will be returned into a standard lymphoedema compression garment, fitted by the research nurse. Thereafter, standard follow up (Bilateral) measurements and checks will be done at 1 month, 3 months, 6 months and 1 year.
  Interventions: Procedure: Lymphaticovenous anastomosis surgery combined with near infrared spectroscopy imaging
- Non-surgical cohort (No Intervention): The main intervention for the non-surgical group largely encompasses limb measurements with perometry and bio-impedance spectroscopy at baseline before a compression garment is applied. The compression garments will be measured and fitted by a trained lymphoedema specialist and will be given the standard advice as is best practice for such patients currently. This cohort will likewise be followed up at 1 month, 3 months, 6 months and 1 year and undergo perometry readings and measurements with comparable collection of data.
  For patients in both surgical and non-surgical groups, the compression garments will be measured and fitted by a trained lymphoedema specialist and they will be given the standard advice as is best practice for such patients currently. For each patient key details of the surgical technique, garment specification, imaging results and perometry/BIS measurements will be recorded on a study specific form for subsequent entry onto the database.

INTERVENTIONS:
Procedure: Lymphaticovenous anastomosis surgery combined with near infrared spectroscopy imaging — Lymphoedema is well recognized as a chronic debilitating disease resulting from an abnormal collection of protein-rich fluid within the subcutaneous tissues of the body. Given the need to identify more effective treatments, more recent advances in super microsurgical techniques have seen the introduction of new procedures, perhaps the most successful of which have involved re-routing the lymphatic fluid by using microsurgery to divert small lymphatic channels into venules in the sub-dermal plane (LVA surgery). This procedure is performed under regional or general anaesthetic as a day-case operation, leaving only a few very short scars in the skin of the arm or leg.
  Arms: Surgical Cohort

SUMMARY:
Lymphoedema is a chronic debilitating disease that can have severe adverse effects on day-to-day life causing great physical and visual discomfort. The clinical presentation is characterised by chronic swelling of limbs, accompanied by localised pain, skin changes and recurrent infections. It is caused by a disruption in lymphatic flow which prevents the normal circulation of interstitial fluid (situated in the spaces between the cells of the body), resulting in swelling of the affected limb. It can be primary (cause unknown) or secondary to a number of causes such as malignancy, trauma, surgery, radiotherapy, infection, or venous disease.

In breast cancer treatment, axillary surgery and radiotherapy significantly damage normal lymphatic drainage of the upper limb, causing lymphoedema in 1-in-5 patients.

There is a growing body of evidence that this chronic and debilitating condition can be better managed through early surgical intervention rather than the current conservative management, which rely on pressure garments and massage. This surgical intervention, lymphaticovenous anastomosis (LVA), joins up a number of the draining lymphatic vessels to correspondingly sized veins on the affected limb using microsurgical techniques. A special dye and camera system is used to facilitate identifying lymph vessels. This creates a new drainage pathway for the lymph fluid around the area of disruption, improving lymphatic flow. Volume reduction is expected and this would be expected to provide quality of life benefits for the patients.

This study seeks to compare the outcomes from both therapies and determine whether LVA surgery can help to improve the physical burden and quality of life for patients affected by lymphoedema. Furthermore, lymphoedema places a substantial burden on NHS services. If this trial is successful, LVA surgery could improve patient outcomes and reduce the overall cost of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients treated with axillary surgery who have developed post-surgical lymphoedema (increase in limb volume by >10% for 1 month or longer)
* Patients must have completed their adjuvant therapy (excluding hormonal/long term Rx)
* Patients must be within 6 months of having developed documented lymphoedema

Exclusion Criteria:

* • Contraindications to the use of the contrast agent (iodine allergy / untreated hypothyroidism)

  * Near infra-red spectroscopy providing insufficient data to guide surgery or evidence of LVA incompatibility (As these patients will be have only just developed lymphoedema, they are by definition very early in the spectrum of disease progression. Thus, the chances of all superficial lymphatics deteriorating to the extent that LVA surgery is not possible is extremely low - <1% we expect).
  * Inability to give informed consent or cooperate with assessment procedures and follow-up because of cognitive or physical impairments
  * Medical co-morbidities increasing the risk of general anaesthetic (significant cardiac / respiratory disease)
  * Recurrent, metastatic or progressive disease, defined by oncology team on basis of clinical assessment or imaging
  * Evidence of pre-existing / primary lymphoedema on clinical history or lymphoscintigraphy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All participants will be having treatment for female breast cancer
Enrollment: 64 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Mean excess volume reduction - compared between two cohorts | 12 months from recruitment
  Primary outcome measure is to evaluate the efficacy of LVA surgery (combined with CGT) by comparison of arm volume measurements across both the surgical and the control group at set time points post-surgery). This will be performed using the mean excess volume reduction (EVR) as a percentage change at 12 months - measured with perometry.

SECONDARY OUTCOMES:
Safety - infection and surgical complications | 12 months from recruitment
  Assess the safety of LVA surgery (supported by PDE imaging guidance) by recording incidence of infection and post-operative complications.
Bio-impedance spectroscopy | 12 months from recruitment
  Compare changes in bio-impedance spectroscopy during the period of the study
Cellulitis | 12 months from recruitment
  Compare the incidence of cellulitis in both groups within the 12-month study period
Quality of life - LYMQOL score | 12 months from recruitment
  Compare longer term Quality of Life (QOL) in both groups using a quality of life assessment tool for lymphoedema of the limbs (LYMQOL) completed by patients. Multiple questions covering function, appearance, symptoms and mood are asked, with a quality of life score for each between 1 and 4. Total score 16 (higher score = poorer quality of life)
Compliance | 12 months from recruitment
  Compliance with use of compression therapy during the study.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Mark Brandon-Grove, Sutton, Surrey
  - Mark Brandon-Grove, London

IPD SHARING:
Plan to Share IPD: No